CLINICAL TRIAL: NCT07111390
Title: A Feasibility Pilot Study of Home-Based Intermittent 60Hz Light Therapy for the Treatment of Depression
Brief Title: Feasibility of Home-Based Intermittent 60Hz Light Therapy for Major Depressive Disorder (MDD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Syntropic Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-00522
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Depression; MDD; Major Depressive Disorder; Major Depressive Episode
Keywords: Brain stimulation; MDD; Depression; Light therapy; Wearable; Neuromodulation; Telehealth
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Home-Based Intermittent Light Therapy (Experimental): Adults with a major depressive episode (MDE) randomized to receive active home-based 60Hz intermittent light therapy, delivered five days per week for three weeks for a total of 15x30-minute daily sessions.
  Interventions: Device: 60Hz Intermittent Light Therapy
- Sham Home-Based Light Therapy (Sham Comparator): Adults with a major depressive episode (MDE) randomized to receive sham home-based light therapy, delivered five days per week for three weeks for a total of 15x30-minute daily sessions.
  Interventions: Device: Sham Light Therapy

INTERVENTIONS:
Device: 60Hz Intermittent Light Therapy — Intermittent 60 Hz flickering white light delivered via a wearable headset.
  Arms: Active Home-Based Intermittent Light Therapy
Device: Sham Light Therapy — Constant white light delivered via a wearable headset.
  Arms: Sham Home-Based Light Therapy

SUMMARY:
This pilot study evaluates the feasibility, safety, and preliminary efficacy of home-based 60Hz intermittent light therapy in adults with a major depressive episode (MDE). Participants will be randomized in a 2:1 ratio to receive either active or sham 60Hz intermittent light stimulation for 30 minutes daily (Monday through Friday) over three weeks. The light is delivered through a wearable headset. Clinical assessments will be conducted remotely at baseline, mid-point, post-treatment, and follow-up to measure changes in depressive symptoms.

DETAILED DESCRIPTION:
This pilot study will evaluate the tolerability, usability, and preliminary impact of a novel wearable device delivering 60Hz intermittent light for treatment of depressive symptoms in adults with MDD. All procedures are conducted remotely.

ELIGIBILITY:
Inclusion Criteria:

* Age between 24 and 65 years (inclusive)*.
* Confirmed diagnosis of Major Depressive Disorder (MDD), based on MINI interview.
* Hamilton Depression Rating Scale (HDRS-17) score ≥17 at screening.
* On a stable dose of antidepressant medication for at least 30 days prior to HDRS-17 screening.
* No evidence of premorbid cognitive impairment, as demonstrated by a standard score >85 on the WRAT-5 Reading Recognition Subtest.
* Confirmed access to a local provider that has primary responsibility for the subjects' clinical care, and who is available for contact in case of increased subject risk due to depressive symptoms.
* Able to provide informed consent and comply with study procedures.
* Access to a quiet space suitable for home-based light stimulation sessions.
* English speaking: All study materials and assessments are only validated in English

Exclusion Criteria:

* Presence of primary neurological or autoimmune disorders.
* Presence of psychiatric comorbidities as determined by the MINI interview (e.g., anxiety disorders, OCD, PTSD, bipolar disorder, psychotic disorder).
* Current or recent diagnosis of alcohol or substance use disorder.
* History of bipolar disorder or any psychotic disorder.
* Clinically significant suicidal ideation or behavior, based on clinician judgment and the Columbia-Suicide Severity Rating Scale (C-SSRS).
* History of seizure disorder or epilepsy.
* History of migraine, tinnitus, or photosensitivity.
* Diagnosis of retinal disease, cataract, or other visual impairments that may interfere with light exposure.
* Regular use of anti-inflammatory drugs or anticoagulants (e.g., clopidogrel).
* Pregnancy and Breastfeeding: Currently pregnant, planning pregnancy during the study period, or breastfeeding

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants who Complete all Scheduled Sessions | Up to Week 3
  Measure of retention; 15 sessions scheduled in total.
Average Percentage of Completed Sessions | Up to Week 3
  Measure of adherence; 15 sessions scheduled in total.
Proportion of Participants who Discontinue due to Adverse Effects | Up to Week 3
  Measure of tolerability.

SECONDARY OUTCOMES:
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) Score | Baseline, Week 3
  The MADRS is a 10-item assessment of depression; each item is rated on a 7-point scale from 0 to 6. The total score is the sum of responses and ranges from 0 to 60; higher scores indicate greater severity of depression.
Change in Hamilton Depression Rating Scale (HDRS-17) Score | Baseline, Week 3
  The HDRS-17 is a 17-item scale assessing the severity of depression. Most items are rated on a 5-point scale (0-4), with some using a 3-point scale (0-2). The total score is the sum of responses and ranges from 0-52; higher scores indicate greater severity of depression.
Change in Patient Health Questionnaire (PHQ-9) Score | Baseline, Week 3
  The PHQ-9 is a 9-item scale assessing the prevalence of depressive symptoms. Each item is rated on a 4-point Likert scale from 0 to 3. The total score is the sum of responses and ranges from 0-27; higher scores indicate greater prevalence of depressive symptoms.
Change in Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR) Score | Baseline, Week 3
  The QIDS-SR is a 15-item scale assessing depressive symptoms over the previous 7 days. Each item is rated on a 4-point Likert scale from 0 to 3. The total score is the sum of responses and ranges from 0-45; higher scores indicate greater prevalence of depressive symptoms.
Change in Work and Social Adjustment Scale (WSAS) Score | Baseline, Week 3
  The WSAS is a 5-item scale assessing the impact of mental health on daily activities. Each item is rated on a 9-point Likert scale from 0 to 8. The total score is the sum of responses and ranges from 0-40; higher scores indicate more severe impairment on daily activities.
Change in Generalized Anxiety Disorder (GAD-7) Score | Baseline, Week 3
  The GAD-7 is a 7-item scale assessing the severity of generalized anxiety disorder. Each item is rated on a scale from 0 to 3. The total score is the sum of responses and ranges from 0-21 with higher scores indicating more severe anxiety.
Post-Study System Usability Questionnaire (PSSUQ) Score | Week 3
  The PSSUQ assesses the overall usability of the intervention; each of the 16 items is rated on a scale from 1-7. The total score is the sum of responses and ranges from 16 to 112; higher scores indicate greater usability of the intervention.
System Usability Scale (SUS) Score | Week 3
  The SUS is a 10-item assessment of the usability of the intervention; the items are rated on a scale from 1-5. The total score is the sum of responses and ranges from 10 to 50; higher scores indicate greater usability of the intervention.
Net Promoter Score (NPS) | Week 3
  The NPS is a single-item questionnaire asking participants how likely they are to recommend the intervention to a colleague. The total score ranges from 1-10; higher scores indicate greater likelihood of promoting the intervention.
Brief Blinding Questionnaire (BBQ) Score | Week 3
  After completing the intervention phase of the study, effectiveness of participant blinding will be assessed using a 3-item questionnaire. The outcome will be scored as the percentage of participants who correctly guess their blinding assignment.
Adverse Events | Week 3
  Incidence of spontaneously reported adverse events during the intervention period. Incidence and type will be reported in the "Adverse Events" section of the results.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppina Pilloni, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the small sample size and risk of re-identification, as well as the exploratory nature of the pilot study.